CLINICAL TRIAL: NCT00677053
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Study of the Safety and Efficacy of TAK-442 in Subjects With Acute Coronary Syndromes
Brief Title: Safety and Efficacy of TAK-442 in Subjects With Acute Coronary Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-442_202; U1111-1112-5867 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Acute Coronary Syndrome
Keywords: Unstable Angina; Myocardial Infarction; Thrombolysis; Anticoagulant; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; Myocardial Infarction | interventions — 1-(1-(3-((6-chloronaphthalen-2-yl)sulfonyl)-2-hydroxypropanoyl)piperidin-4-yl)tetrahydropyrimidin-2(1H)-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- TAK-442 10 mg BID (Experimental): Added with standard care for recurrent ischemic events.
  Interventions: Drug: TAK-442
- TAK-442 20 mg BID (Experimental): Added with standard care for recurrent ischemic events
  Interventions: Drug: TAK-442
- TAK-442 40 mg QD (Experimental): Added with standard care for recurrent ischemic events
  Interventions: Drug: TAK-442
- TAK-442 40 mg BID (Experimental): Added with standard care for recurrent ischemic events
  Interventions: Drug: TAK-442
- TAK-442 80 mg QD (Experimental): Added with standard care for recurrent ischemic events
  Interventions: Drug: TAK-442
- TAK-442 80 mg BID (Experimental): Added with standard care for recurrent ischemic events
  Interventions: Drug: TAK-442
- TAK-442 160 mg QD (Experimental): Added with standard care for recurrent ischemic events
  Interventions: Drug: TAK-442
- TAK-442 120 mg BID (Experimental): Added with standard care for recurrent ischemic events
  Interventions: Drug: TAK-442
- Placebo (Placebo Comparator): Added with standard care for recurrent ischemic events
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-442 — Stage I: TAK-442 10 mg, capsules, orally, twice daily and standard care for recurrent ischemic events for up to 24 weeks.
  Arms: TAK-442 10 mg BID
Drug: TAK-442 — Stage I: TAK-442 20 mg, capsules, orally, twice daily and standard care for recurrent ischemic events for up to 24 weeks.
  Arms: TAK-442 20 mg BID
Drug: TAK-442 — Stage I: TAK-442 40 mg, capsules, orally, once daily and standard care for recurrent ischemic events for up to 24 weeks.
  Arms: TAK-442 40 mg QD
Drug: TAK-442 — Stage II: TAK-442 40 mg, capsules, orally, twice daily and standard care for recurrent ischemic events for up to 24 weeks.
  Arms: TAK-442 40 mg BID
Drug: TAK-442 — Stage II: TAK-442 80 mg, capsules, orally, once daily and standard care for recurrent ischemic events for up to 24 weeks.
  Arms: TAK-442 80 mg QD
Drug: TAK-442 — Stage II: TAK-442 80 mg, capsules, orally, twice daily and standard care for recurrent ischemic events for up to 24 weeks.
  Arms: TAK-442 80 mg BID
Drug: TAK-442 — Stage III: TAK-442 160 mg, capsules, orally, once daily and standard care for recurrent ischemic events for up to 24 weeks.
  Arms: TAK-442 160 mg QD
Drug: TAK-442 — Stage III: TAK-442 120 mg, capsules, orally, twice daily and standard care for recurrent ischemic events for up to 24 weeks.
  Arms: TAK-442 120 mg BID
Drug: Placebo — Stages I, II & III: TAK-442 placebo-matching capsules, orally, twice daily and standard care for recurrent ischemic events for up to 24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability of multiple doses of TAK-442once daily, (QD) or twice daily (BID), in subjects with acute coronary syndrome (unstable angina, myocardial infarction).

DETAILED DESCRIPTION:
Acute coronary syndrome, including myocardial infarction with or without ST-segment elevation and stable or unstable angina, is acknowledged to represent collectively a major global healthcare problem. Despite existing treatments, the rates of patient mortality, myocardial infarction and hospital readmissions during follow-up remain very high.

Due to its critical role in propagating the blood coagulation cascade, activated factor X now is considered to be a major therapeutic target in the development of novel antithrombotic therapy by blocking thrombin generation and attenuating the formation of fibrin. Therefore, activated factor X inhibitors, exhibiting either indirect or direct modes of action, are among the novel agents under investigation in the treatment of acute coronary syndrome.

This study will evaluate the safety and tolerability of TAK-442 compared with placebo in post-acute coronary syndrome subjects who are also receiving standard antiplatelet and other cardiovascular therapy.

Individuals who want to participate in this study will be required to provide written informed consent. Study participation is anticipated to be approximately 3.5 months. Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, physical examinations, electrocardiograms and bilateral venogram.

ELIGIBILITY:
Inclusion Criteria:

* Has been hospitalized for acute coronary syndrome
* Is able to initiate study drug if:

  * The index event occurred within the past 7 days (the date of initial hospitalization will be utilized for the date on which the index event occurred), and
  * The final acute medical or cardiac procedural intervention for the treatment of acute coronary syndrome was last administered or performed at least 36 hours before administration of the first dose of study drug.
* Has at least 1 of the following additional ischemic risk factors:

  * Previous myocardial infarction.
  * The index event was an anterior myocardial infarction.
  * Presence of multivessel coronary disease
  * Left bundle branch block.
  * Left ventricular ejection fraction less than 40% at any time during hospitalization for the index event.
  * Killip class greater than or equal to II at any time during hospitalization for the index event.
  * History of symptomatic congestive heart failure
  * History of ischemic stroke or transient ischemic attack.
  * Presence of peripheral arterial obstructive disease.
  * Diabetes mellitus requiring medical therapy to maintain glycemic control.
  * Current smoker
  * Moderate renal impairment
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* Has low body weight greater than 50 kg.
* Has severe hypertension.
* Has a known bleeding/clotting disorder.
* Has acute pericarditis.
* Has a history of intracranial or intraocular bleeding.
* Has a history of gastrointestinal bleeding or gastric or duodenal ulceration.
* Has a history of ischemic stroke or transient ischemic attack.
* Has had major surgery, including coronary artery bypass graft or has undergone non-major laparoscopic surgery or non-major minimally invasive surgery, within 2 weeks prior to Randomization.
* Has a history of cancer that has not been in remission for at least 5 years.
* Has a condition for which long-term anticoagulation therapy is indicated or requires ongoing use of other excluded medications.
* Has severe renal dysfunction.
* Has anemia or thrombocytopenia that has not resolved prior to Randomization.
* Has alanine aminotransferase or total bilirubin levels greater than 2 times the upper limit of normal, active liver disease or jaundice.
* Has a history of illicit drug use or excessive alcohol intake.
* Has any other serious disease or condition that would compromise subject safety, increase the risk of bleeding, or make it difficult to successfully manage and follow the subject according to the protocol.
* Has received TAK-442 in a previous clinical study or as a therapeutic agent.
* Has a history of hypersensitivity or allergies to other fXa inhibitors.
* Has received any investigational compound within 30 days prior to Screening or is currently participating in another study which entails the administration of an investigational or marketed drug, supplement or intervention including, but not limited to diet, exercise, lifestyle or invasive procedure.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * azole antifungal agents
  * cyclosporine
  * clarithromycin
  * HIV protease inhibitors
  * nefazodone
  * ritonavir
  * quinidine
  * amiodarone
  * verapamil

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2753 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Major Bleeding Events defined by the Thrombolysis in Myocardial Infarction Scale. | On Occurrence (Up to 24 weeks)

SECONDARY OUTCOMES:
Composite of Cardiovascular Mortality, non-fatal Myocardial Infarction, non-fatal Stroke, or Myocardial Ischemia requiring hospitalization. | Week 24
Cardiovascular Mortality. | Week 24.
Non-fatal Myocardial Infarction. | Week 24.
Non-fatal Stroke. | Week 24.
Myocardial Ischemia requiring hospitalization. | Week 24.
All-cause Mortality. | Week 24.
Hemorrhagic Mortality. | Week 24.
Composite of Cardiovascular death, non-fatal Myocardial Infarction, or Myocardial Ischemia requiring hospitalization. | Week 24.
Composite of Cardiovascular death, non-fatal Myocardial Infarction, or non-fatal Stroke. | Week 24.
Hospitalization for Heart Failure. | Week 24.
Incidence of minor bleeding events defined by the Thrombolysis in Myocardial Infarction Scale. | On Occurrence (Up to 24 weeks).
Incidence of minimal bleeding events defined by the Thrombolysis in Myocardial Infarction Scale. | On Occurrence (Up to 24 weeks).
Incidence of major, clinically significant non-major bleeding AND minor bleeding events as defined by the Secondary Bleeding Scale | On Occurrence (Up to 24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director Clinical Science, Study Director — Takeda
Locations (103):
- United States (15):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Pensecola, Florida
  - West Des Moines, Iowa
  - Salisbury, Maryland
  - Minneapolis, Minnesota
  - Cherry Hill, New Jersey
  - Toledo, Ohio
  - Sayre, Pennsylvania
  - Houston, Texas
  - Victoria, Texas
  - Layton, Utah
  - Roanoke, Virginia
- Buenos Aires, Argentina
- Belgium (3):
  - Bonheiden
  - Genk
  - Liège
- Brazil (2):
  - Porto Algere
  - Recife
- Bulgaria (9):
  - Haskovo
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Rousse
  - Silistra
  - Sofia
  - Stara Zagora
  - Varna
- Canada (5):
  - Greater Sudbury, Ontario
  - Toronto, Ontario
  - Chilliwack
  - Saint-Charles-Borromée
  - Vancouver
- Chile (2):
  - Santiago
  - Temuco
- Tallinn, Estonia
- Germany (2):
  - Bad Nauheim
  - Langen
- Hungary (7):
  - Budapest
  - Debrecen
  - Nyíregyháza
  - Szeged
  - Székesfehérvár
  - Szolnok
  - Zalaegerszeg
- India (14):
  - Ahmedabad
  - Bikaner
  - Calicut
  - Indore
  - Jaipur
  - Mangaluru
  - Mumbai
  - Nagpur
  - New Delhi
  - Pune
  - Shimoga
  - Thrissur
  - Trivandrum
  - Vadodara
- Netherlands (5):
  - Amsterdam
  - Hardenberg
  - Hoorn
  - The Hague
  - Tilburg
- Peru (2):
  - Arequipa
  - Lima
- Romania (8):
  - Bacau
  - Baia Mare
  - Brasov
  - Brăila
  - Bucharest
  - Cluj-Napoca
  - Suceava
  - Târgovişte
- Russia (12):
  - Barnaul
  - Kemerovo
  - Krasnoyarsk
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Samara
  - Saratov
  - Tomsk
  - Tyumen
  - Voronezh
  - Yaroslavl
- Serbia (2):
  - Kamenica
  - Sremska
- South Africa (8):
  - Bloemfontein
  - CapeTown
  - Goodwood
  - Johannesburg
  - Parow
  - Pinelands
  - Pretoria
  - Randburg
- South Korea (4):
  - Busan
  - Daegu
  - Jeonrabukdo
  - Seoul
- Airdrie, North Lanarkshire, United Kingdom